CLINICAL TRIAL: NCT06913335
Title: Optimizing Hemostasis in Laparoscopic Ovarian Cystectomy: A Comparison Between Electrosurgical Energy and Hemostatic Sealants.
Brief Title: Comparison Between Electrosurgical Energy and Hemostatic Sealants on Hemostasis in Laparoscopic Ovarian Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Aya Yasser Fawzy, resident, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-504
Record Dates: First submitted 2025-03-23; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- electrosurgical energy group (Active Comparator): in this group electrosurgical energy will be used to control bleeding
  Interventions: Procedure: laparoscopic ovarian cystectomy using electrosurgical energy
- Hemostatic Sealant group (Active Comparator): in this group Hemostatic Sealant will be used to control bleeding
  Interventions: Procedure: laparoscopic ovarian cystectomy using hemostatic sealant

INTERVENTIONS:
Procedure: laparoscopic ovarian cystectomy using hemostatic sealant — * A small incision will be made on the ovarian surface using laparoscopic scissors.
  * Nontraumatic grasping forceps will be used to dissect the cyst capsule away from the soft tissue of the ovary.
  * The cyst will be removed intact to avoid spillage of its contents. If rupture occurs, the peritoneal cavity will be irrigated thoroughly.
  * After the removal of the cyst, the ovarian bed should be inspected for bleeding, and if there is minimal bleeding, using of electrocautery should be avoided to minimize thermal damage to the ovary.
  * The hemostatic sealant as Surgicel original, Surgicel Fibrillar (ETHICON, USA) which is an absorbable hemostat (oxidized regenerated cellulose) will be applied directly to the bleeding surface 1:5sheets of hemostat will be used.
  Arms: Hemostatic Sealant group
Procedure: laparoscopic ovarian cystectomy using electrosurgical energy — A small incision will be made on the ovarian surface using laparoscopic scissors.
  * Nontraumatic grasping forceps will be used to dissect the cyst capsule away from the soft tissue of the ovary.
  * The cyst will be removed intact to avoid spillage of its contents. If rupture occurs, the peritoneal cavity will be irrigated thoroughly.
  * After the removal of the cyst, the ovarian bed should be inspected for bleeding, and if there is minimal bleeding, using of electrocautery should be avoided to minimize thermal damage to the ovary In the electrosurgical energy using group the hemostasis method will be different and will be achieved using electrosurgical energy.
  * After the cyst removal and cyst bed examination, any bleeding will be carefully coagulated using bipolar electrosurgical energy
  * Minimal energy will be applied for short durations to reduce collateral thermal
  Arms: electrosurgical energy group

SUMMARY:
The aim of this study is to compare between the effect of using electrosurgical energy and hemostatic sealant for hemostasis in laparoscopic cystectomy for ovarian cysts.

DETAILED DESCRIPTION:
Ovarian cysts are common in women during childbearing period. Most cysts are normal functional cysts that typically resolve spontaneously and need no treatment. However, pathologic cysts such as endometriomas and dermoid may require surgical intervention.( For women of childbearing age with symptomatic ovarian cysts, laparoscopic cystectomy is the first-line surgical treatment for ovarian cysts because it has many advantages, including the benefits of ovarian-sparing surgery (with continued hormonal support and preservation of future fertility) and of minimally invasive surgery (including small incisions, quick recovery, and less pain).

Laparoscopic ovarian cystectomy is the treatment of choice for benign ovarian tumors in the young, including mature cystic teratomas, endometriomas, and serous or mucinous cystadenomas. One of the greatest challenge during the surgery is stopping bleeding from the rest ovarian tissue.

Electrosurgical energy is a commonly used technique to cut off bleeding from the remaining ovarian tissue during laparoscopic ovarian cystectomy, but it can increase time of operation , increase the risk of complications, and if used excessively, it can damage the soft tissues of the ovaries, and interfere with fertility .

Electrosurgical units can be divided into two major types: monopolar and bipolar, monopolar system refers to current flow from one active electrode through the patient, who is entirely included in the circuit, and exists via dispersive electrode to the generator, but its usage can cause collateral injuries and thermal necrosis at the point of contact.

In bipolar units, both active and return electrodes are housed within the same instrument; so, the current flows only through the tissue between the two blades of the electrode and return to the generator without passing through the whole body.

Bipolar energy is safer than monopolar energy in terms of the risk of postoperative adhesions and the risk of over treatment that can lead to ovarian failure and also provide a significant postoperative resumption of the spontaneous ovulation and pregnancy.

On the other hand, other hemostatic strategies have been investigated such as hemostatic sealants, which create a seal when applied to bleeding tissues. This process causes platelets to clump together and initiates the clotting cascade, obstructing blood flow.

Other studies, including randomized controlled trials, have consistently demonstrated that hemostatic sealants are effective in stopping bleeding and reducing blood loss at many surgical sites. This empirical evidence demonstrates the potential of a hemostatic sealant as an effective alternative to electrosurgical energy, particularly in surgical situations that require strong hemostasis, such as laparoscopic ovarian cystectomy.

Ovarian reserve is defined as the size and number of the ovarian follicle pools at any given time. Alternatively, it can be defined as the total ovarian follicle pool which is equal to the quiescent (primordial) follicles plus growing follicles. This reproductive potential is determined by the quiescent primordial follicles that can develop into primary, antral, and ovulating follicles. It can be estimated by several methods and the level of serum anti-Mullerian hormone (AMH) is considered one of the best endocrine markers .

AMH is formed by the granulosa cells of active follicles (primary follicles, preantral follicles and small antral follicles) but not by quiescent primordial follicles. AMH regulates the process of follicle formation by controlling the number of primordial follicles that initiate the maturation process, thus preventing the exhaustion of the quiescent follicles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Women with unilateral or bilateral benign ovarian cyst provisionally diagnosed by ultrasound and normal tumor markers.
* Women fit for laparoscopic surgery

Exclusion Criteria:

* Pregnant women.
* Postmenopausal women.
* Premenarchal girls.
* Women with a history of recent pelvic or abdominal radiotherapy.
* Women with serious concurrent systemic disorders.
* Known ovarian malignancy provisionally diagnosed by ultrasound (US) or tumor markers.
* Women with coagulopathy or bleeding disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study will be the hemostasis time | Day 1
  The primary outcome of this study will be the hemostasis time

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No